CLINICAL TRIAL: NCT00787878
Title: Comparison of Safety in Small for Gestational Age (SGA) Subjects Treated With Norditropin® (Somatropin) 5 Years Ago With Untreated SGA Subjects and With Normal Average for Gestational Age (AGA) Subjects
Brief Title: Long Term Metabolic Safety of Norditropin® Treatment of Small for Gestational Age (SGA) Subjects
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: GHLIQUID-1975
Record Dates: First submitted 2008-11-07; First posted 2008-11-10 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Foetal Growth Problem; Small for Gestational Age
MeSH Terms: interventions — Human Growth Hormone

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- A
  Interventions: Drug: somatropin
- B
  Interventions: Drug: No treatment given
- C
  Interventions: Drug: No treatment given

INTERVENTIONS:
Drug: somatropin — SGA previously treated with Norditropin®
  Other Names: GHLIQUID
  Groups: A
Drug: No treatment given — Untreated SGA
  Groups: B
Drug: No treatment given — AGA (Average gestational age)
  Groups: C

SUMMARY:
The study is conducted in Europe. The primary aim of this observational study is to compare the insulin sensitivity in small for gestational age (SGA) subjects treated with Norditropin® with untreated small for gestational age (SGA) subjects and with average for gestational age (AGA) subjects.

ELIGIBILITY:
Inclusion Criteria:

* Norditropin® treated small for gestational age (SGA) group: Treated with Norditropin® for at least three years in the IUGR-1 or IUGR-2 trials
* Untreated small for gestational age (SGA) group: Birth length and/or weight less than -2 SDS for gestational age
* Average gestational age (AGA) group: Birth length and/or weight larger than -2 SDS for gestational age

Exclusion Criteria:

* Growth hormone deficiency defined as a peak growth hormone (GH) less than 20 mU/l
* Insulin like growth (IGF)-1 level less than -2 SDS
* Receipt of any investigational drug within four weeks prior to the trial

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: GH treated SGA and controls of non-treated SGA and AGA
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2009-02; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | Index 5 years after end of GH treatment compared to controls

SECONDARY OUTCOMES:
Disposition index, glucose effectiveness and acute insulin response compared to controls | 5 years after end of Norditropin treatment

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Rotterdam, Netherlands

REFERENCES:
- [Result] van Dijk M, Bannink EM, van Pareren YK, Mulder PG, Hokken-Koelega AC. Risk factors for diabetes mellitus type 2 and metabolic syndrome are comparable for previously growth hormone-treated young adults born small for gestational age (sga) and untreated short SGA controls. J Clin Endocrinol Metab. 2007 Jan;92(1):160-5. doi: 10.1210/jc.2006-1073. Epub 2006 Oct 24. PMID 17062774
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com